CLINICAL TRIAL: NCT05517941
Title: Effect of Active Cycle Breathing Technique Along With Incentive Spirometer on COVID19 Patient
Acronym: COVID19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator. alshaymaa shaaban abd el-azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003416
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Corona Virus Infection
Keywords: active cycle breathing; incentive spirometer; covid19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: active cycle breathing and incentive spirometer
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active cycle breathing exercise (Experimental): patients will receive Active cycle of breathing techniques daily for 2 weeks
  Interventions: Other: active cycle breathing
- incentive spirometer (Experimental): patients will receive incentive spirometer and active cycle breathing daily for 2 weeks
  Interventions: Other: active cycle breathing; Other: incentive spirometer

INTERVENTIONS:
Other: active cycle breathing — The active cycle breathing technique will involve three steps: breathing control, thoracic expansion exercise, and forced expiration technique, In breathing control, the patient will sit comfortably in a chair and breathe at a normal rate and depth using the lower chest. In the thoracic expansion exercise, the physical therapist rested his/her hands on the patient's epigastrium and guided the patient's breathing so that they breathed at a slow and deep rate using the lower chest, then held their breath for 2 s and fully exhaled; this was repeated two or three times, then the patient returned to breathing control. For the forced expiration technique, the physical therapist asked the patient to inhale deeply while simultaneously contracting the abdominal muscle and keeping the mouth and throat open. They then held their breath for 2 s, followed by vigorous exhalation
Other: incentive spirometer — Incentive spirometry is accomplished by using a device that provides feedback when the patient inhales at a predetermined flow and sustains the inflation for at least 5 seconds. The patient is instructed to hold the spirometer in an upright position, exhale normally, and then place the lips tightly around the mouthpiece. The next step is a slow inhalation to raise the ball (flow-oriented) or the piston/ plate (volume-oriented) in the chamber to the set target. At maximum inhalation, the mouthpiece is removed, followed by a breath-hold and normal exhalation.
  Arms: incentive spirometer

SUMMARY:
this study will be conducted to investigate the effect of Active Cycle Breathing Technique and incentive spirometer on COVID19 patient

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a new coronavirus that emerged in 2019 and causes coronavirus disease 2019 (COVID-19).Individuals with COVID-19 can present with an influenza-like illness and respiratory tract infection demonstrating fever (89%),cough (68%), fatigue (38%), sputum production (34%) and/or shortness of breath (19%). The spectrum of disease severity ranges from asymptomatic infection or mild upper respiratory tract illness through to severe viral pneumonia with respiratory failure and/or death. Current reports estimate that 80% of cases are asymptomatic or mild; 15% of cases are severe (infection requiring oxygen); and 5% are critical, requiring ventilation and life support. Based on emerging data, individuals at the highest risk of developing severe COVID-19 disease requiring hospitalization and/or ICU support are those who are older, male, have at least one co-existing comorbidity, elevated D-dimer levels, and/or lymphocytopenia. Active cycle breathing techniques (ACBT) is a cycle of techniques consisting of breathing control, lower thoracic expansion exercises and the forced expiration technique modifiable to individual patients. It assists bronchial clearance by enhancing mucociliary clearance whilst reducing adverse effects such as hypoxemia or increased airflow obstruction. Incentive spirometry (IS) is a type of deep breathing exercise that is widely used for lung expansion and the prevention of pulmonary complications in children, adults, and the elderly. IS is used to encourage the patient to inhale to lung capacity through maximal inspiration aided with visual feedback. These maneuvers increase transpulmonary pressure and therefore increase chest-wall volume.one hundred patients will be allocated randomly to two groups; one group will receive active cycle breathing with an incentive spirometer and the other will receive active cycle breathing

ELIGIBILITY:
Inclusion Criteria:

* Ages from 45-75 years old
* COVID-19 patients with SpO2 > 85
* oxygen face Mask or a reservoir mask

Exclusion Criteria:

* Mechanically ventilated,
* Cancer,
* Chronic respiratory disease (defined as asthma or chronic obstructive pulmonary disease),
* End-stage renal disease,
* Liver disease (defined as compensated/decompensated liver cirrhosis),
* Chronic neurological disease (defined as previous neurological disease),
* Chronic cardiovascular disease,
* Active smoker

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
arterial blood gas | up to two weeks
  arterial blood gas analysis will be measured using arterial blood sample

SECONDARY OUTCOMES:
C-reactive protein | up to two weeks
  C-reactive protein will be measured by blood sample analysis
Oxygen saturation | up to two weeks
  SpO2 will be measure by pulse oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- El sheikh zayed Al nahyan hospital, Giza, Egypt